CLINICAL TRIAL: NCT00086944
Title: A Phase I/II Study of G3139 (Genasense) in Combination With RICE Chemotherapy in Relapsed B-Cell Non-Hodgkin's Lymphoma
Brief Title: Oblimersen, Rituximab and Combination Chemotherapy in Treating Patients With Relapsed or Refractory Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02600; 12975A; N01CM62201 (NIH); CDR0000371904 (Registry Identifier: PDQ (Physician data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — oblimersen; Rituximab; Ifosfamide; indolepropanol phosphate; Carboplatin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim

ARMS (1):
- Treatment (genase, combination chemotherapy) (Experimental): See detailed description.
  Interventions: Biological: oblimersen sodium; Biological: rituximab; Drug: ifosfamide; Drug: carboplatin; Drug: etoposide; Biological: filgrastim; Biological: pegfilgrastim; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Biological: pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of oblimersen when given together with rituximab and combination chemotherapy and to see how well they work in treating patients with relapsed or refractory aggressive non-Hodgkin's lymphoma. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as ifosfamide, carboplatin, and etoposide, work in different ways to stop cancer cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of chemotherapy by making cancer cells more sensitive to the drugs

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of oblimersen when given in combination with rituximab, ifosfamide, carboplatin, and etoposide in patients with relapsed or refractory aggressive B-cell non-Hodgkin's lymphoma.

II. Determine the safety and toxicity of this regimen in these patients. III. Determine the complete and partial response rate in patients treated with this regimen.

SECONDARY OBJECTIVES:

I. Determine the duration of response, overall survival, and time to progression in patients treated with this regimen.

II. Determine the effect of this regimen on hematopoietic stem cell kinetics and yield from these patients.

OUTLINE: This is a multicenter, phase I, dose-escalation study of oblimersen followed by a phase II study.

Phase I: Patients receive GRICE comprising oblimersen IV continuously on days 1-5, rituximab IV, ifosfamide IV continuously over 24 hours, and carboplatin IV over 1 hour on day 4, and etoposide IV over 30 minutes once daily on days 4-6. Treatment repeats every 14 days for 3 courses. Patients also receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 7 and continuing until blood counts recover OR one dose of pegfilgrastim SC on day 7 of courses 1 and 2. For course 3, all patients receive G-CSF SC twice daily beginning on day 7 and continuing until stem cell collection is complete. Patients with responding disease who are not eligible for autologous SCT may receive up to 8 total courses of GRICE or 2 additional courses beyond maximal response. Patients with responding disease to GRICE who are eligible for autologous SCT are removed from the study and undergo autologous SCT off study. Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Phase II: Patients receive oblimersen at the MTD determined in phase I and rituximab, ifosfamide, carboplatin, and etoposide followed by G-CSF or pegfilgrastim as in phase I. In both phases, treatment continues in the absence of disease progression, unacceptable toxicity, or the patient becomes a candidate for autologous SCT. Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed aggressive B-cell non-Hodgkin's lymphoma

  * Any 1 one of the following histological subtypes for phase I:

    * Grade 3 follicular center lymphoma
    * Diffuse large B-cell lymphoma
    * Transformed follicular lymphoma
    * Mantle cell lymphoma
    * Primary mediastinal B-cell lymphoma
  * Any 1 of the following histological subtypes for phase II:

    * Diffuse large B-cell lymphoma
    * Transformed follicular lymphoma
    * Primary mediastinal B-cell lymphoma
* Measurable disease

  * At least 1 bidimensionally measurable lesion ≥ 10 mm in longest diameter by CT scan, MRI, x-ray, or clinical exam
* Relapsed disease after 1, and only 1, prior anthracycline-based chemotherapy regimen
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* Absolute neutrophil count ≥ 1,000/mm^3*
* Platelet count ≥ 100,000/mm^3*
* Bilirubin normal**
* AST and ALT ≤ 2.5 times upper limit of normal
* PT and PTT normal
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to oblimersen or other study drugs
* No currently active second malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix

  * Must have completed any prior therapy for a second malignancy and is considered to be at < 30% risk of relapse
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* Prior rituximab allowed
* No other concurrent immunotherapy
* See Disease Characteristics
* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy
* No concurrent hormonal therapy
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent therapeutic radiotherapy
* At least 4 weeks since prior surgery
* No prior oblimersen or other antisense oligonucleotide therapy
* No other concurrent anticancer agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-05; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Toxicity graded using the NCI CTCAE version 3.0 | Up to 3 years
Complete and partial response rate according to the International Workshop Criteria | Up to 3 years

SECONDARY OUTCOMES:
Duration of response | From the time measurement criteria are met for CR/CRu/PR until the first date that PD is objectively documented, assessed up to 3 years
Overall survival | From the first day of therapy to the date of death, assessed up to 3 years
Time to progression | From the first day of treatment until the date PD or death is first reported, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Smith, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States